CLINICAL TRIAL: NCT02262767
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo Controlled, Single Ascending Dose Study To Investigate The Safety, Tolerability, And Pharmacokinetics Of Pf 06649751 Co-administered With Trimethobenzamide Hydrochloride In Healthy Volunteers
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of PF-06649751 Co-administered With Trimethobenzamide Hydrochloride in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7601007; 2014-003631-19 (EudraCT Number)
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Phase 1, Randomized, Double Blind, Placebo-Controlled, Single-Dose Escalation, Safety, Tolerability, Pharmacokinetic, PF-06649751, Trimethobenzamide
MeSH Terms: interventions — trimethobenzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Ascending Doses Cohort 1 (Experimental): Single doses, given by oral solution, starting at 0.75 mg up to a possible maximum of 3.0 mg. The subject will have been fasted for 10 hours prior to the single dose. For each dosing period, 3 subjects will be given a placebo as a comparator while 6 are given active dose. The subjects will be given concomitant trimethobenzamide hydrochloride for the 3 weeks that the subject is in the CRU. For each of the three periods, subjects will be crossed-over from placebo or PF-06649751. Each PF-06649751 dose is separated by one week.
  Interventions: Drug: PF-06649751; Drug: Trimethobenzamide Hydrochloride
- Single Ascending Doses Cohort 2 (Experimental): Single doses, given by oral solution, starting at 4.5 mg up to a possible maximum of 9.0 mg. The subject will have been fasted for 10 hours prior to the single dose. For each dosing period, 3 subjects will be given a placebo as a comparator while 6 are given active dose. The subjects will be given concomitant trimethobenzamide hydrochloride for the 3 weeks that the subject is in the CRU. For each of the three periods, subjects will be crossed-over from placebo or PF-06649751. Each PF-06649751 dose is separated by one week.
  Interventions: Drug: PF-06649751; Drug: Trimethobenzamide Hydrochloride

INTERVENTIONS:
Drug: PF-06649751 — Experimental Pfizer compound.
Drug: Trimethobenzamide Hydrochloride — Trimethobenzamide Hydrochloride is indicated for the treatment of postoperative nausea and vomiting and for nausea associated with gastroenteritis.
  Other Names: Tigan

SUMMARY:
This study will test the hypothesis that PF-06649751 with continuous co-administration of trimethobenzamide hydrochloride (TMB) with will be safe and well tolerated. Single doses of PF-06649751 will be tested in this study, starting at a low dose and escalating to a dose projected to be under the current limits for drug concentration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication (whichever is longer).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 0 - 4 weeks
  Counts of participants who have treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to PF-06649751 will be assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category will be counted once within the category.
Supine and standing vital sign measurements | 0 - 4 weeks
  Measurement of blood pressure and pulse rate.
Electrocardiogram (ECG) | 0 - 4 weeks
  Measurement of standard 12-lead ECG, single or triplicate
Number of Participants With Laboratory Test Values of Potential Clinical Importance | 0 - 4 weeks
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1
  Maximum plasma concentration
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Day 1 - 5
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Area Under the Curve From Time Zero to Extrapolated Infinite Time AUCinf | Day 1 - 5
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0 - t) plus AUC (t - inf).
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1
Plasma Decay Half-Life (t1/2) | Day 1 - 5
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | Day 1 - 5
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | Day 1 - 5
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Constantino Kantaridis, MD, Principal Investigator — Pfizer
Locations (2):
- Belgium (2):
  - Belgium Pfizer Clinical Research Unit, Brussels
  - Pfizer Clinical Research Unit, Brussels